CLINICAL TRIAL: NCT01592578
Title: A Randomized Controlled Trial of Ligation Versus Ligation Plus Sclerotherapy in Addition to Cyanoacrylate in Patients With Gastroesophageal Varices
Brief Title: The Research of the Evaluation of Clinical Procedures in Gastroesophageal Varices in Patients With Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, department of Gastroenterology, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSY-CJ-2012
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2012-05

CONDITIONS: Gastroesophageal Varice
Keywords: gastroesophgeal variceal bleeding; liver cirrhosis; portal hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Ligation; Cyanoacrylates; Sclerotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ligation and Cyanoacrylate Group (Active Comparator)
  Interventions: Procedure: Ligation and Cyanoacrylate
- Ligation plus Sclerotherapy and Cyanoacrylate Group (Experimental)
  Interventions: Procedure: Ligation plus Sclerotherapy and Cyanoacrylate Group

INTERVENTIONS:
Procedure: Ligation and Cyanoacrylate — Patients will be treated with ligation for esophageal varices and cyanoacrylate for gastric varices when necessary.
  Arms: Ligation and Cyanoacrylate Group
Procedure: Ligation plus Sclerotherapy and Cyanoacrylate Group — Patients will receive sclerotherapy after first ligation for esophageal varices and cyanoacrylate for gastric varices when necessary
  Arms: Ligation plus Sclerotherapy and Cyanoacrylate Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of two different endoscopic treatment in gastroesophageal varices in patients with liver cirrhosis: ligation versus ligation plus sclerotherapy in addition to cyanoacrylates

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding, which often results from portal hypertention, is known as one of the most frequent death causes of patients with liver cirrhosis. When a patient has bleeding episode, it's very likely that he/she will develop another one in the future. Endoscopic treatments such as ligation, sclerotherapy or cyanocrylates are proved to decrease the risk of re-bleeding. The purpose of this study is to evaluate the efficacy of two different endoscopic treatments in patients who have both gastric and esophageal varices with liver cirrhosis: In addition to cyanoacrylates, ligation versus ligation plus sclerotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with portal hypertension caused by liver cirrhosis who presented with an acute or recent episode of gastroesophageal variceal bleeding and have previously received endoscopic treatments of ligation and cyanoacrylate. Diagnosis of liver cirrhosis or mixed cirrhosis was based on results of liver biopsy or biochemical tests and liver imaging by ultrasonography.
* The extent of the varices range from Moderate to Severe.
* The age of the patients range from 18 to 72 years old.

Exclusion Criteria:

* Patients who had other causes for portal hypertention(CTPV,Budd-Chiari syndrome,etc.)
* Patients with severe systemic disease (renal failure, heart failure,carcinoma other than liver cancer,etc.)
* Patients who had contraindications for ligation,sclerotherapy or cyanoacrylate.
* Patients who have previously received shunt or devascularization operation,TIPS.
* Patients who had portosystemic shunt according to the results of CT scan.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of variceal hemorrhage | Participants will be followed for up to 6 months starting from the date of randomization.
  recurrence rate of variceal hemorrhage

SECONDARY OUTCOMES:
eradication rate of the gastroesophageal varices | Participants will be followed for up to 6 months starting from the date of randomization.Eradication of the gastroesophageal varices will be measured according to the results of endoscopy at the end of the 6 months.
  We intend to set eradication rate of the gastroesophageal varices as one of our secondary outcomes. Participants will be followed for up to 6 months starting from the date of randomization.Eradication of the gastroesophageal varices will be measured according to the results of endoscopy at the end of the 6 months.
recurrence rate of the gastroesophageal varices | Participants will be followed for up to 6 months starting from the date of randomization.Recurrence rate of the gastroesophageal varices will be measured according to the results of endoscopy at the end of the 6 months.
  We intend to set recurrence rate of gastroesophageal varices as one of our secondary outcomes. Participants will be followed for up to 6 months starting from the date of randomization.Recurrence rate of the gastroesophageal varices will be measured according to the results of endoscopy at the end of the 6 months.
mortality rate during the follow-up period | Participants will be followed for up to 6 months starting from the date of randomization.
  mortality rate during the follow-up period
incidence rate of complications associated with endoscopic treatments | Participants will be followed for up to 6 months starting from the date of randomization.
  We intend to set incidence rate of complications associated with endoscopic treatments,to be specific,which include trasient fever, transient dysphagia, transient arrhythmias, ulceration, perforation, stricture, rebleeding, aspiration pneumonia, sepsis, peritonitis and chest pain. Participants will be followed for up to 6 months starting from the date of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen J, Zeng XQ, Ma LL, Li B, Tseng YJ, Lian JJ, Gao H, Wang J, Luo TC, Chen SY. Randomized controlled trial comparing endoscopic ligation with or without sclerotherapy for secondary prophylaxis of variceal bleeding. Eur J Gastroenterol Hepatol. 2016 Jan;28(1):95-100. doi: 10.1097/MEG.0000000000000499. PMID 26517621